CLINICAL TRIAL: NCT00420576
Title: A Randomized, Double-Blind, Multiple-Dose Escalation Study of the Effect of Danggui Buxue Tang on Symptomatic Postmenopausal Hong Kong Chinese Women (Continuation of a Completed Study Using the Same Formula)
Brief Title: Dose Finding Study of Danggui Buxue Tang (Herbal Formula)on the Treatment of Menopausal Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: The Institute of Chinese Medicine, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ICM/CTS/05/336
Record Dates: First submitted 2007-01-09; First posted 2007-01-11 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2007-01

CONDITIONS: Postmenopausal
Keywords: Post-menopausal; Traditional Chinese Medicine; Randomized
MeSH Terms: interventions — danggui buxue decoction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): Low Dose Danggui Buxue Tang (1.5g)
  Interventions: Drug: DBT-Danggui Buxue Tang
- 2 (Experimental): Middle Dose Danggui Buxue Tang(3g)
  Interventions: Drug: DBT-Danggui Buxue Tang
- 3 (Experimental): High Dose Danggui Buxue Tang (6g)
  Interventions: Drug: DBT-Danggui Buxue Tang

INTERVENTIONS:
Drug: DBT-Danggui Buxue Tang — Herbal Combination of Danggui (Radix Angelicae Sinensis) and Huangqi (Radix Astragali)in granules form, in 3 different dosage 6g/3g/1.5g, once time per day for 3 Months treatment
  Other Names: Danggui Buxue Tang

SUMMARY:
Main purpose of the study is to look for an optimal dose for the treatment of menopausal symptoms with the Chinese Herbal Medicines containing Dang Gui and Huang Qi.

DETAILED DESCRIPTION:
The menopause implies the permanent cessation of menstrual bleeding. In western medicine, this is associated either with the spontaneous failure of normal ovarian function, or it may also result from surgical removal of the ovaries or as a consequence of chemotherapy or radiotherapy. In western medicine, the usual treatment of the menopause is the use of oestrogen replacement therapy. However, treatment with oestrogen may result in unwanted side effects such as breast soreness and nausea. In addition, the long-term safety of oestrogen treatment has not been established. Oestrogen is therefore a valuable treatment for the menopause, but it is not without side effects. It remains to be seen whether Chinese Medicine as described in this proposal can prove to be an effective, safe and well tolerated treatment for the menopause. Dang Gui (Radix Angelicae Sinensis) is one Chinese herb that is recommended for the treatment of menopausal symptoms. Huang Qi is also used in the treatment of the menopausal symptoms to tonify Qi. We have now shown a beneficial effect of Danggui Buxue Tang on vasomotor symptoms in postmenopausal Chinese women (Re: CREC Ref. No. CRE-2002.152-T). However, we could not show a difference in the reduction in severity of symptoms between Danggui Buxue Tang and placebo. We now wish to confirm our initial findings, and we hope to obtain more reliable data by (1) only including women who have never used any type of treatment for their menopause and (2) by recruiting women who have more severe symptoms of the menopause.

Chinese Herbal Medicines containing Dang Gui and Huang Qi have been used for many years to treat menopausal women. There are few data on possible adverse effects of treatment with Chinese Herbal Medicine containing Dang Gui as well as Huang Qi..

The objective of present study is to investigate the dose response relationship to assess an optimal dose suitable for clinical use. The trial will be designed as a multiple-dose escalation clinical trial to obtain accurate information on the efficacy and safety when used for menopausal women. Since previous study has already confirmed that the dose used was efficacious, the main purpose of the study is to look for an optimal dose for the treatment of menopausal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Follicle stimulating hormone (FSH), luteinizing hormone (LH), oestradiol in the menopausal range (FSH>18 IU/L, LH>12.6 IU/L, and E2< 361 pmol/l)
* Patients with amenorrhoea for more than 12 months
* Never received treatment for menopausal symptoms
* Never received menopausal hormone therapy
* Reporting a minimum of 21 hot flushes per week at the time of entry into the study

Exclusion Criteria:

* Patients with a history of using Chinese medicine or other therapies which may affect the outcome within 8 weeks
* Patients who in the judgment of the investigator will be unable to comply with protocol requirements.
* Patients with significant gastrointestinal, renal, hepatic, bronchopulmonary, neurological, cardiovascular, breast or endometrial carcinoma, or allergic diseases;
* Patients with uncontrolled hypertension,
* Patients with undiagnosed vaginal bleeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
the changes in severity and frequency of hot flushes and sweats (menopausal symptoms) | 5 Months

SECONDARY OUTCOMES:
the changes of score on the Menopause specific quality of life | 5 Months
the changes in values of various markers of risk for cardiovascular disease | 5 Months

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Haines, FPOGS, Principal Investigator — Department of Obstetrics & Gynaecology, CUHK
Locations (1):
- Department of Obstetrics & Gynaecology, CUHK, Prince of Wales Hospital, Hong Kong, China

REFERENCES:
- [Background] Hagstad A, Janson PO. The epidemiology of climacteric symptoms. Acta Obstet Gynecol Scand Suppl. 1986;134:59-65. doi: 10.3109/00016348609157052. PMID 3468732
- [Background] Schneider HP, Gallagher JC. Moderation of the daily dose of HRT: benefits for patients. Maturitas. 1999 Nov;33 Suppl 1:S25-9. doi: 10.1016/s0378-5122(99)00060-2. PMID 10661612
- [Background] Au GK. Evaluation of the benefits and risks of hormone replacement therapy. Hong Kong Med J. 2000 Dec;6(4):381-9. PMID 11177160
- [Background] Blumel JE, Castelo-Branco C, Binfa L, Gramegna G, Tacla X, Aracena B, Cumsille MA, Sanjuan A. Quality of life after the menopause: a population study. Maturitas. 2000 Jan 15;34(1):17-23. doi: 10.1016/s0378-5122(99)00081-x. PMID 10687878
- [Background] Hall G, Pripp U, Schenck-Gustafsson K, Landgren BM. Long-term effects of hormone replacement therapy on symptoms of angina pectoris, quality of life and compliance in women with coronary artery disease. Maturitas. 1998 Jan 12;28(3):235-42. doi: 10.1016/s0378-5122(97)00080-7. PMID 9571599
- [Background] Zhu DP. Dong quai. Am J Chin Med. 1987;15(3-4):117-25. doi: 10.1142/S0192415X87000151. PMID 3425569
- [Background] Davis SR, Briganti EM, Chen RQ, Dalais FS, Bailey M, Burger HG. The effects of Chinese medicinal herbs on postmenopausal vasomotor symptoms of Australian women. A randomised controlled trial. Med J Aust. 2001 Jan 15;174(2):68-71. doi: 10.5694/j.1326-5377.2001.tb143156.x. PMID 11245505
- [Background] Fugh-Berman A. Herb-drug interactions. Lancet. 2000 Jan 8;355(9198):134-8. doi: 10.1016/S0140-6736(99)06457-0. PMID 10675182
- [Background] Chung TK, Yip SK, Lam P, Chang AM, Haines CJ. A randomized, double-blind, placebo-controlled, crossover study on the effect of oral oestradiol on acute menopausal symptoms. Maturitas. 1996 Oct;25(2):115-23. doi: 10.1016/0378-5122(96)01050-x. PMID 8905602